CLINICAL TRIAL: NCT03916016
Title: Sí Texas HOPE: Enhanced Integrated Behavioral Health Model for Uninsured Patients
Brief Title: Sí Texas Hope Family Health Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources in Action, Inc. (Other)
Collaborators: Methodist Healthcare Ministries of South Texas, Inc. (Unknown); Social Innovation Fund (Unknown)
Responsible Party: Principal Investigator, Karen Errichetti, Director, Research and Evaluation, Health Resources in Action, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100002
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Chronic Disease; Hypertension; Diabetes; Hypercholesterolemia; Depression; Obesity
Keywords: Integrated Behavioral Health; Integrated Care; Volunteer Clinic
MeSH Terms: conditions — Chronic Disease; Hypertension; Diabetes Mellitus; Hypercholesterolemia; Depression; Obesity

STUDY DESIGN:
Intervention Model Description: Treatment group participants were randomized to receive enhanced integrated behavioral health care. Control group participants received care as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group received enhanced integrated behavioral health care.
  Interventions: Behavioral: Enhanced Integrated Behavioral Health Care
- Control Group (Active Comparator): The control group received care as usual only.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Enhanced Integrated Behavioral Health Care — The intervention involved moving from HFHC's previous collaborative model, where medical and behavioral providers worked with each other episodically, to a more fully integrated collaborative care model with care coordination, shared treatment plans, shared service provision, and shared record keeping. To achieve this enhanced level of integration, HFHC changed its current primary care workflow to include a behavioral health specialist who conducted assessments, provided initial counseling (individual or group), and coordinated referrals to care management and/or community-based health services.
  Arms: Intervention Group
Behavioral: Usual Care — A collaborative model where medical and behavioral providers worked with each other episodically
  Arms: Control Group

SUMMARY:
This study evaluated whether uninsured patients living at or below 200% of the federal poverty level who received enhanced, culturally-relevant, integrated behavioral health services were more likely to improve health outcomes after 12 months compared to similar patients receiving usual care from Hope Family Health Center (HFHC), a charitable community clinic. The study employed a randomized control trial (RCT) design where intervention participants receiving integrated care at HFHC were compared to control participants receiving usual care at HFHC. Patients were placed in each group using simple random assignment. Demographic and health outcome data were collected from intervention and control participants at baseline. Health outcome data were subsequently collected at 6-month and 12-month follow-up points.

DETAILED DESCRIPTION:
This study evaluated whether uninsured patients living at or below 200% of the federal poverty level who received enhanced, culturally-relevant, integrated behavioral health services were more likely to improve health outcomes after 12 months compared to similar patients receiving usual care from Hope Family Health Center (HFHC), a charitable community clinic. The study employed a randomized control trial (RCT) design where intervention participants receiving integrated care at HFHC were compared to control participants receiving usual care at HFHC. Patients were placed in each group using simple random assignment. Demographic and health outcome data were collected from intervention and control participants at baseline. Health outcome data were subsequently collected at 6-month and 12-month follow-up points. The primary outcomes of interest were systolic and diastolic blood pressure and depressive symptoms. Additional secondary outcomes of interest were HbA1c and BMI. These outcomes were analyzed as continuous variables using linear regression with backward model selection. Longitudinal analyses were also conducted using a likelihood-based approach to general linear mixed models. The participants (1) resided in Cameron, Hidalgo, Willacy, or Starr County, (2) were eligible to receive behavioral health services from HFHC (e.g., uninsured, living at or below 200% of the federal poverty level, residence in HFHC's service area), and (3) had a diagnosis of hypertension (blood pressure of 140/90 mm Hg or higher) and/or obesity (body mass index of 30.0 or higher) and/or poorly controlled diabetes (HbA1c over 6.8) and/or moderate depression (score of 10 or above on PHQ-9).

ELIGIBILITY:
Inclusion Criteria:

* Reside in Cameron, Hidalgo, Starr, or Willacy County
* Were eligible to receive behavioral health services from HFHC (e.g., uninsured, living at or below 200% of the federal poverty level, residence in HFHC's service area)
* Have a diagnosis of one or more chronic conditions:
* Hypertension (blood pressure of 140/90 mmHg or higher)
* Obesity (body mass index of 30.0 or higher)
* Poorly controlled diabetes (HbA1c over 6.8%)
* Moderate depression (score of 10 or above on PHQ-9)

Exclusion Criteria:

* Not actively suicidal at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | One year
  Blood pressure was measured as a continuous variable (systolic and diastolic) in millimeters of mercury (mmHg).

SECONDARY OUTCOMES:
Body mass index | One year
  Height and weight were measured at baseline, and body mass index was calculated.
Depressive Symptoms | One year
  Score calculated based on responses to the Patient Health Questionnaire-9. The PHQ-9 has a total possible score of 27. Each of the nine questions is assigned a value of 0, 1, 2, or 3. The total score is the sum of individual questions' scores. The PHQ-9 scoring criteria is categorized as minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27) depression.
Blood glucose concentration | One year
  Blood glucose concentration was measured via blood test for HbA1c as a continuous variable

IPD SHARING:
Plan to Share IPD: No